CLINICAL TRIAL: NCT06699277
Title: Diagnostic Accuracy of Chest Ultrasonography Vs. Chest X-ray in the Evaluation of Chest Trauma: a Comparative Study Using CT As the Gold Standard.
Brief Title: Chest Ultrasound Versus Chest X-ray with Ct As Gold Standard At Trauma Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Omar elmokhtar Abdelaziz khalaf Mohamed Ali, Resident, Assiut University
Other Study IDs: Chest ultrasound vs X-ray
Record Dates: First submitted 2024-11-19; First posted 2024-11-21 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Pneumothorax At Trauma Patients

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this observational study is to learn about the predictive value of the chest ultrasound in detection of pneumothorax at chest trauma patients.

The main question it aims to answer is:

How does the performance of the chest ultrasound compare to chest X-ray in predicting pneumothorax in chest trauma patients in Egypt? Participants are patients with different ages Isolated blunt chest trauma patients admitted to the emergency department during the study period.

DETAILED DESCRIPTION:
Chest trauma is a leading cause of morbidity and mortality, with timely and accurate diagnosis essential for effective treatment. While chest X-ray (CXR) has traditionally been the first-line imaging modality in emergency settings due to its availability and ease of use, it has limitations, particularly in detecting subtle or occult injuries like pneumothorax, haemothorax, rib fractures, and pulmonary contusions, especially in trauma patients positioned supine. Overuse of CXR can also lead to increased costs, radiation exposure, and emergency department overcrowding.

Ultrasound has emerged as an alternative, with multiple studies showing that chest ultrasonography (CUS) is highly sensitive and specific for detecting traumatic intrathoracic injuries, including pneumothorax. This systematic review and meta-analysis aimed to assess the diagnostic accuracy of CUS compared to CXR. While CT scans remain the gold standard for diagnosing thoracic trauma due to their superior accuracy, they expose patients to significant radiation and should be used judiciously. Although CXR is a fast and accessible option in emergencies, it may miss critical injuries, highlighting the importance of balancing diagnostic accuracy with patient safety and resource management in trauma care.

The primary aim of this study is to evaluate and compare the diagnostic accuracy of chest ultrasonography (sonar) versus chest X-ray (CXR) in the detection of thoracic injuries in patients presenting with chest trauma, using computed tomography (CT) as the reference standard.

ELIGIBILITY:
Inclusion Criteria:

* patients with different ages.
* both genders.
* Patients presenting with isolated blunt chest trauma.
* Patients who are hemodynamically stable and can undergo imaging studies (Ultrasonography, CXR, and CT).
* Patients who provide informed consent (or proxy consent if the patient incapacitated).

Exclusion Criteria:

* Hemodynamically unstable patients requiring immediate surgical intervention.
* Patients with contraindications to CT imaging (e.g., severe renal impairment without access to alternative contrast agents).
* Pregnant patients (due to radiation exposure from CT).
* Patients with previous thoracic surgery or pre-existing significant thoracic abnormalities that could interfere with imaging interpretation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Blunt chest trauma patients admitted to emergency departments in Assuit and Suez Canal University Hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of chest ultrasonography compared to chest X-ray in the Evaluation of Chest Trauma patients. | Hour 3 after patient arrival to ER.
  To evaluate and compare the diagnostic accuracy of chest ultrasonography (sonar) versus chest X-ray (CXR) in the detection of thoracic injuries in patients presenting with chest trauma, using computed tomography (CT) as the reference standard.

IPD SHARING:
Plan to Share IPD: No